CLINICAL TRIAL: NCT06163989
Title: The Protective Impact of TheaLoz Duo Eyedrop on the Ocular Surface in Hand-Held Console and Computer Game Users
Brief Title: Protecting the Eyes of Gamers With Lubricating Eyedrops
Acronym: PROTEGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aston University (Other)
Responsible Party: Principal Investigator, Jeremy Chiang, Postdoctoral Research Associate, Aston University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HLS21135
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Dry Eye Syndromes; Computer Vision Syndrome
Keywords: Lubricating eyedrop; Artificial tears; Ocular surface
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either the active treatment (TheaLoz Duo) or control condition (no eyedrops) at the first visit. The cross-over will occur one month following the first phase, followed by another month when the participant will be assessed again at the final visit.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TheaLoz Duo in first month, crossover to control condition in second month (Experimental): The TheaLoz Duo eyedrop will be prescribed and used by the participant for 1 month. At the second visit 1 month later, the participant will return the TheaLoz Duo eyedrop bottle, and no eyedrops will be prescribed, and the participant monitored following 1 month. At the third and final visit 1 month later, the participant will return for a follow-up visit.
  Interventions: Drug: TheaLoz Duo Eyedrop
- Control condition in first month, crossover to TheaLoz Duo in second month (Active Comparator): No eyedrops will be prescribed and the participant monitored for 1 month. At the second visit 1 month later, the participant will return and be prescribed TheaLoz Duo eyedrop and used by the participant for another 1 month. At the third and final visit 1 month later, the participant will return the TheaLoz Duo eyedrop bottle and complete the study visits.
  Interventions: Drug: TheaLoz Duo Eyedrop

INTERVENTIONS:
Drug: TheaLoz Duo Eyedrop — TheaLoz Duo lubricating eyedrop contains 3.0% trehalose and 0.15% sodium hyaluronate as active ingredients and will be used by participants everyday to instill 1 drop, 4 times a day in both eyes.
  Other Names: Treatment Eyedrop

SUMMARY:
The excessive use of screens particularly amongst digital gamers can adversely impact the health of the surface of the eyes with symptoms and signs of surface damage. While strategies including limiting screen time exist, these may be ineffective given the widespread rise of digital device use and gaming culture in the modern era. There is limited evidence for the protective effect of lubricating eyedrops on the ocular surface for handheld console and computer gamers.

The aim of this study is to investigate the protective effect of a lubricating eyedrop (TheaLoz Duo) on the surface of the eyes in handheld console and computer gamers. The main question it aims to answer is whether TheaLoz Duo could protect the surface of the eyes from dessication and alleviate symptoms of dry eye disease in handheld console and computer gamers.

Participants will receive either the lubricating eyedrop first for 1 month, followed by a control condition (no eyedrops) for another month, or the other way round. Participants will attend 3 visits in total, each separated by 1 month apart. During each visit, routine clinical assessments of the front of the eye will be conducted. Subsequent findings from this timely study will help improve care of the surface of the eyes for a growing population of gamers worldwide.

DETAILED DESCRIPTION:
This study will be a randomized, outcome assessor-masked, cross-over clinical study to assess the potential impact of TheaLoz Duo lubricating eyedrop on symptoms and signs of dry eye disease in handheld console and computer gamers. All visits will be conducted at the Aston Dry Eye Clinic in Aston University, Birmingham, United Kingdom.

ELIGIBILITY:
Inclusion criteria:

* Individuals with dryness symptoms as assessed with the Ocular Surface Disease Index (OSDI score ≥ 13).
* Individuals who play handheld console and computer-based games ≥ 2 hours everyday on average
* Individuals who are comfortable and competent at using smartphone applications
* Age ≥ 18 years, male or female
* Able to provide written consent in English
* Able to instil the treatment lubricating eyedrop on their own, and return any provided eyedrop bottle to the researcher used at the end of the treatment
* Able to attend multiple visits (3 visits over 2 months)

Exclusion criteria:

* Pregnancy
* Use of any topical ocular medical eyedrops or lubricants in the 1 week prior to starting the study or during the study period. Those who are using existing lubricating eyedrops and are interested in participating will be required to stop their lubricating eyedrops for 1 week prior to commencing the study
* History of ocular surgery, trauma or infections in the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Ocular Surface Disease Index scores to the First Follow-Up 1 Month After Baseline | Baseline to 1 month after baseline
  Validated questionnaire for assessing dry eye symptom severity and impact. Scores range from 0 indicating no dry eye symptoms to 100 with severe dry eye symptoms and impact (Schiffman et al, 2000).
Change from First Follow-Up in Ocular Surface Disease Index scores to the Second Follow-Up 1 Month After the First Follow-Up | First follow-up to 1 month after the first follow-up
  Validated questionnaire for assessing dry eye symptom severity and impact. Scores range from 0 indicating no dry eye symptoms to 100 with severe dry eye symptoms and impact (Schiffman et al, 2000).

SECONDARY OUTCOMES:
Change from Baseline in Computer Vision Syndrome Questionnaire scores to the First Follow-Up 1 Month After Baseline | Baseline to 1 month after baseline
  Validated questionnaire for assessing the severity and frequency of eye strain when using a computer. The scores range from 0 to 32 (Seguí Mdel et al, 2015).
Change from First Follow-Up in Computer Vision Syndrome Questionnaire scores to the Second Follow-Up 1 Month After the First Follow-Up | First follow-up to 1 month after the first follow-up
  Validated questionnaire for assessing the severity and frequency of eye strain when using a computer. The scores range from 0 to 32 (Seguí Mdel et al, 2015).
Change from Baseline in Visual Acuity to the First Follow-Up 1 Month After Baseline | Baseline to 1 month after baseline
  Subjective measure of visual acuity using Logarithm of the Minimum Angle Resolution (logMAR) scoring, ranging from -0.30 which signify the ability to be able to resolve the smallest letters, to 1.00 which signify the ability to resolve only the largest letters.
Change from First Follow-Up in Visual Acuity to the Second Follow-Up 1 Month After the First Follow-Up | First follow-up to 1 month after the first follow-up
  Subjective measure of visual acuity using Logarithm of the Minimum Angle Resolution (logMAR) scoring, ranging from -0.30 which signify the ability to be able to resolve the smallest letters, to 1.00 which signify the ability to resolve only the largest letters.
Change from Baseline in Tear Meniscus Height to the First Follow-Up 1 Month After Baseline | Baseline to 1 month after baseline
  Measure of the volume of tears in mm using the Oculus Keratograph 5M instrument. An average of 3 measurements is obtained.
Change from First Follow-Up in Tear Meniscus Height to the Second Follow-Up 1 Month After the First Follow-Up | First follow-up to 1 month after the first follow-up
  Measure of the volume of tears in mm using the Oculus Keratograph 5M instrument. An average of 3 measurements is obtained.
Change from Baseline in Lipid Layer Pattern to the First Follow-Up 1 Month After Baseline | Baseline to 1 month after baseline
  Subjective grading of the appearance of the lipid layer pattern as a surrogate measure of its thickness using the Oculus Keratograph 5M instrument. This ranges from Grade 1 indicating very thin lipid layer to Grade 6 indicating very thick lipid layer.
Change from First Follow-Up in Lipid Layer Pattern to the Second Follow-Up 1 Month After the First Follow-Up | First follow-up to 1 month after the first follow-up
  Subjective grading of the appearance of the lipid layer pattern as a surrogate measure of its thickness using the Oculus Keratograph 5M instrument. This ranges from Grade 1 indicating very thin lipid layer to Grade 6 indicating very thick lipid layer.
Change from Baseline in Bulbar Conjunctival Hyperaemia to the First Follow-Up 1 Month After Baseline | Baseline to 1 month after baseline
  Automated objective grading of the bulbar conjunctival redness using the Oculus Keratograph 5M instrument. This ranges from Grade 0 indicating no redness to Grade 4 indicating substantial redness.
Change from First Follow-Up in Bulbar Conjunctival Hyperaemia to the Second Follow-Up 1 Month After the First Follow-Up | First follow-up to 1 month after the first follow-up
  Automated objective grading of the bulbar conjunctival redness using the Oculus Keratograph 5M instrument. This ranges from Grade 0 indicating no redness to Grade 4 indicating substantial redness.
Change from Baseline in Blink Rate to the First Follow-Up 1 Month After Baseline | Baseline to 1 month after baseline
  Manual subjective count of the number of blinks using the Oculus Keratograph 5M instrument.
Change from First Follow-Up in Blink Rate to the Second Follow-Up 1 Month After the First Follow-Up | First follow-up to 1 month after the first follow-up
  Manual subjective count of the number of blinks using the Oculus Keratograph 5M instrument.
Change from Baseline in Fluorescein Corneal Staining to the First Follow-Up 1 Month After Baseline | Baseline to 1 month after baseline
  Subjective grading of the amount of corneal staining using fluorescein instillation, cobalt blue light illumination and the Oxford grading scale. This ranges from 0 with no staining to 5 with intense staining.
Change from First Follow-Up in Fluorescein Corneal Staining to the Second Follow-Up 1 Month After the First Follow-Up | First follow-up to 1 month after the first follow-up
  Subjective grading of the amount of corneal staining using fluorescein instillation, cobalt blue light illumination and the Oxford grading scale. This ranges from 0 with no staining to 5 with intense staining.
Change from Baseline in Lissamine Green Bulbar Conjunctival Staining to the First Follow-Up 1 Month After Baseline | Baseline to 1 month after baseline
  Subjective grading of the amount of bulbar conjunctival staining using lissamine green instillation, white light illumination and the Oxford grading scale. This ranges from 0 with no staining to 5 with intense staining.
Change from First Follow-Up in Lissamine Green Bulbar Conjunctival Staining to the Second Follow-Up 1 Month After the First Follow-Up | First follow-up to 1 month after the first follow-up
  Subjective grading of the amount of bulbar conjunctival staining using lissamine green instillation, white light illumination and the Oxford grading scale. This ranges from 0 with no staining to 5 with intense staining.
Change from Baseline in Lissamine Green Lid Wiper Epitheliopathy to the First Follow-Up 1 Month After Baseline | Baseline to 1 month after baseline
  Subjective grading of the amount of lid wiper epitheliopathy using lissamine green instillation and white light illumination. This grading ranges from 0 with no lid wiper epitheliopathy to 4 with severe lid wiper epitheliopathy
Change from First Follow-Up in Lissamine Green Lid Wiper Epitheliopathy to the Second Follow-Up 1 Month After the First Follow-Up | First follow-up to 1 month after the first follow-up
  Subjective grading of the amount of lid wiper epitheliopathy using lissamine green instillation and white light illumination. This grading ranges from 0 with no lid wiper epitheliopathy to 4 with severe lid wiper epitheliopathy
Change from Baseline in Meibography Meiboscore to the First Follow-Up 1 Month After Baseline | Baseline to 1 month after baseline
  Subjective grading of the amount of Meibomian gland loss using infrared imaging and the Pult meiboscore. This grading ranges from 0 with no gland loss to 4 with severe gland loss (Pult and Reide-Pult, 2013).
Change from First Follow-Up in Meibography Meiboscore to the Second Follow-Up 1 Month After the First Follow-Up | First follow-up to 1 month after the first follow-up
  Subjective grading of the amount of Meibomian gland loss using infrared imaging and the Pult meiboscore. This grading ranges from 0 with no gland loss to 4 with severe gland loss (Pult and Reide-Pult, 2013).
Number of Participants with Dry Eye Disease at Baseline | At baseline
  The number of participants diagnosed with dry eye disease according to established clinical diagnostic criteria (Wolffsohn et al, 2017).
Number of Participants with Dry Eye Disease at First Follow-Up | At first follow-up 1 month after baseline
  The number of participants diagnosed with dry eye disease according to established clinical diagnostic criteria (Wolffsohn et al, 2017).
Number of Participants with Dry Eye Disease at SecondFollow-Up | At second follow-up 1 month after first follow-up
  The number of participants diagnosed with dry eye disease according to established clinical diagnostic criteria (Wolffsohn et al, 2017).

CONTACTS AND LOCATIONS:
Overall Officials: James S Wolffsohn, PhD, Study Director — Aston University
Locations (1):
- School of Optometry, Aston University, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The investigators are planning to deposit deidentified datasets in a publicly and freely available data repository site.
Time Frame: Data will be available at the end of the study before publication of the findings in a peer-reviewed journal.
Access Criteria: The dataset will be publicly and freely available.

REFERENCES:
- [Background] Wolffsohn JS, Arita R, Chalmers R, Djalilian A, Dogru M, Dumbleton K, Gupta PK, Karpecki P, Lazreg S, Pult H, Sullivan BD, Tomlinson A, Tong L, Villani E, Yoon KC, Jones L, Craig JP. TFOS DEWS II Diagnostic Methodology report. Ocul Surf. 2017 Jul;15(3):539-574. doi: 10.1016/j.jtos.2017.05.001. Epub 2017 Jul 20. PMID 28736342
- [Background] Schiffman RM, Christianson MD, Jacobsen G, Hirsch JD, Reis BL. Reliability and validity of the Ocular Surface Disease Index. Arch Ophthalmol. 2000 May;118(5):615-21. doi: 10.1001/archopht.118.5.615. PMID 10815152
- [Background] Pult H, Riede-Pult B. Comparison of subjective grading and objective assessment in meibography. Cont Lens Anterior Eye. 2013 Feb;36(1):22-7. doi: 10.1016/j.clae.2012.10.074. Epub 2012 Oct 27. PMID 23108007
- [Background] Segui Mdel M, Cabrero-Garcia J, Crespo A, Verdu J, Ronda E. A reliable and valid questionnaire was developed to measure computer vision syndrome at the workplace. J Clin Epidemiol. 2015 Jun;68(6):662-73. doi: 10.1016/j.jclinepi.2015.01.015. Epub 2015 Jan 28. PMID 25744132